CLINICAL TRIAL: NCT04446143
Title: Effects of Mindfulness Meditation on Patients' Satisfaction During Urodynamic Study.
Brief Title: Effects on Mindfulness Meditation on Patient's Satisfaction During Urodynamic Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5200230
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Personal Satisfaction
Keywords: meditation, urodynamics, satisfaction, pain, anxiety
MeSH Terms: conditions — Personal Satisfaction; Pain; Anxiety Disorders | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Subject randomization will use permutated blocks and assignments in concealed consecutively numbered envelops. Those in the mindfulness medication group will listen to an audio-taped mediation, which takes 10 mins to complete, where as the control group will be seated in a quiet empty room where they wait for 10 min.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application of mindfulness meditation prior to UDS (Other): Those in the mindfulness medication group will listen to an audio-taped mediation, which takes 10 mins to complete.
  Interventions: Behavioral: Mindfulness meditation
- No meditation prior to UDS (Active Comparator): The control group will be seated in a quiet empty room where they wait for 10 min.
  Interventions: Behavioral: Mindfulness meditation

INTERVENTIONS:
Behavioral: Mindfulness meditation — Mindfulness meditation

SUMMARY:
The purpose of this investigator-initiated study is to evaluate if mindfulness-based stress reduction (MBSR) will improve satisfaction and reduce anxiety during a urodynamic study (UDS).

DETAILED DESCRIPTION:
Urodynamic studies (UDS) are used to measure the functionality of the bladder and urethra to be able to evaluate lower urinary tract symptoms (LUTS). UDS consists of catheterization, uroflow and cystometrogram. Intravesical, vaginal or rectal transducer placements, and placement of perineal electrodes are part of the study protocol. During the study the bladder will be filled slowly with sterile fluid and the patient will be asked about sensation of filling. At the end of the study the patient will be asked to void.

Although beneficial for diagnosis of underlying LUTS, UDS maybe associated with heightened patient anxiety and feeling of discomfort. In a recently published pilot study, it was shown that a mindfulness-based stress reduction (MBSR) protocol may help improve a patient's emotional health and perception of UDS. To validate the findings from this previous study, the current study aims to implement a MBSR protocol in a randomized prospective study. Patients scheduled for UDS will be randomized into two groups. One group will listen to mindfulness meditation prior to the UDS and the other group won't.

All patients will complete validated questionnaires to assess their satisfaction, anxiety and pain level as well as lower urinary tract symptoms before and after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Female and male patients between ages 18 and 99 with clinical indication for UDS ordered by treating physician

Exclusion Criteria:

* None English speakers will be recruited for this study.
* Pregnancy
* Prioners

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All genders and gender-identities (phenotype, genotype) are eligible for this study.
Enrollment: 60 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Satisfaction during the urodynamic study testing | 1 year
  Likert scale will measure satisfaction with urodynamics in both groups. The scale ranges are: very dissatisfied=0, dissatisfied=1, somehow satisfied=2, satisfied=3, very satisfied=4), with 0 as the worse outcome.

SECONDARY OUTCOMES:
Self evaluation of anxiety and comfort level | 1 year
  The State-Trait Anxiety Inventory (STAI 6) score will be obtained before and after the study. It measures stress and anxiety. It ranges from: not al all=1, somewhat=2, moderately so=3, very much so=4), with 4 as the worse outcome.
Pain level | 1 year
  The visualised analog pain score (VAS) will be obtained before and after the study. It measure the degree of pain and a range between 0-10 (0=no pain et all and 10=worst pain ever), with 10 as the worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Staack, Principal Investigator — Loma Linda Univ Health
Locations (1):
- Loma Linda University Faculty Medical Offices, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Uberoi P, Smitherman A, Aden J, Park G, Jellison F. Incorporation of Mindfulness Exercises to Reduce Anxiety During Urodynamic Testing: A Randomized Single-Blind Controlled Pilot Trial. J Altern Complement Med. 2020 Jan;26(1):74-75. doi: 10.1089/acm.2018.0447. Epub 2019 Sep 25. No abstract available. PMID 31553223